CLINICAL TRIAL: NCT03975244
Title: Effects of Exercise on Body Composition, Cardiovascular Risk Factors and Surgery Complications in Bariatric Patients
Brief Title: Semi-supervised Exercise Program Before Bariatric Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital General Universitario Elche (Other)
Responsible Party: Principal Investigator, Jaime Ruiz-Tovar, MD, PhD, Department of Surgery, Hospital General Universitario Elche
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRJC-19_Ex.Bar
Record Dates: First submitted 2019-05-30; First posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-05

CONDITIONS: Morbid Obesity; Exercise; Bariatric Surgery
MeSH Terms: conditions — Obesity, Morbid; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): Three months of semi-supervised exercise program in patients awaiting bariatric surgery. Body composition, cardiovascular risk factors, physical fitness, physical activity levels and quality of life will be assessed before and at the end of the study. In addition, surgery time, hospital length of stay and operative complications also will be evaluated.
  Interventions: Behavioral: Exercise program
- Control group (No Intervention): The control group only will perform the evaluations of the study.

INTERVENTIONS:
Behavioral: Exercise program — Twelve-week of semi-supervised exercise program. The exercise program will combine resistance and endurance training. Both the volume and intensity of training will start at moderate intensity, and progressively be increased at higher volumes and intensities.
  Other Names: Exercise program in patients awaiting bariatric surgery.
  Arms: Exercise group

SUMMARY:
Background: Patients awaiting bariatric surgery, apart from suffering higher BMI, show a large number of comorbidities and a low physical fitness. These factors are associated with a longer surgery time, a longer hospital stay and a greater number of operative complications. To reduce these disadvantages, a nutritional intervention is performed to reduce total weight and the comorbidities associated with obesity prior to surgery. However, the prescription of an exercise program, which can be an effective tool to improve these factors, is not usually part of the usual care of these patients.

Objective: To know the effects of a semi-supervised exercise program on body composition, cardiovascular risk factors and operative complications in bariatric patients.

Methods: Approximately 3 months before surgery, 60 patients awaiting bariatric surgery will be recruited. Patients will be randomized into two groups: a) an experimental group (n = 30); b) a control group (n = 30). The experimental group will perform a semi-supervised exercise program, while the control group will only perform the corresponding evaluations. Both groups will be assessed for body composition, cardiovascular risk factors, physical condition, quality of life and physical activity levels at the beginning and at the end of the intervention. In addition, surgery time, hospital length of stay and operative complications will be evaluated in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-55 years.
* All patients awaiting bariatric surgery.

Exclusion Criteria:

* Patients with chronic respiratory diseases
* Patients with cardiovascular diseases
* Inability to perform exercise

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in body composition - Body mass index | Baseline and 3 months, between 8:00 AM and 9:00 AM.
  Bioimpedance analysis will be used for establishing body weight and body composition. This variables will be evaluated between 8:00 and 9:00 A.M., after at least 8 hours of fasting, with an empty bladder. Body mass index will be calculated dividing weight in kilograms by squared height in meters. Therefore, body mass index will be expressed as kg·m-2.
Change in glucose and HbA1c levels. | Baseline and 3 months, between 8:00 AM and 10:00 AM.
  Blood samples will be taken after a 12 h of overnight fast. Exercise will be forbidden 48 h before the test.
Change in total cholesterol, HDL cholesterol and LDL cholesterol levels. | Baseline and 3 months, between 8:00 AM and 10:00 AM.
  Blood samples will be taken after a 12 h of overnight fast. Exercise will be forbidden 48 h before the test.
Change in systolic and diastolic blood pressure. | Baseline and 3 months, between 8:00 AM and 9:00 AM.
  Systolic and Diastolic Blood pressure will be measured according to established recommendations.
Complications rates | Day 30 after surgery.
  All the complications suffered by patients will be recorded.
Length of stay. | Day 15 after surgery.
  The number of days at hospital after bariatric surgery will be recorded.
Change in handgrip strength | Baseline and 3 months, between 5:00 PM and 8:00 PM.
  Strength levels will be assessed using a hand dynamometer.

SECONDARY OUTCOMES:
Change in physical activity levels. | Baseline and 3 months, seven days.
  Levels of physical activity will be measured recording the physical activity performed for 7 days using an accelerometer.
Change in health-related quality of life: sf-36 questionnaire. | Baseline and 3 months.
  The Spanish version of Short Form Health Survey 36 (SF-36) will be used for knowing changes in quality of life. This questionnaire uses 8 scales to evaluate physical health (4 scales: Physical Function, Role Physical, Bodily Pain, General Health) and mental health (4 scales: Vitality, Social functioning, Role Emotional, and Mental Health). The scores of these scales are transformed into values between 0-100 points, where highest scores are related to better function. These 8 scales are grouped into two summary components (physical summary component; mental summary component) which will be calculated according to the reference values of the Spanish population, with a mean of 50 and standard deviation of 10.population.
Change in waist and hip circumference. | Baseline and 3 months, between 8:00 AM and 9:00 AM.
  Waist and hip circumference will be measured in centimeters, using established recommendations.